CLINICAL TRIAL: NCT03714373
Title: An Open-Label, Long-Term Safety and Efficacy Evaluation of Diazoxide Choline Extended-Release Tablets in Participants With Prader-Willi Syndrome With a Double-Blind, Placebo-Controlled, Randomized Withdrawal Period
Brief Title: Open-Label Extension Study of DCCR in PWS Followed by Double-Blind, Placebo-Controlled, Randomized Withdrawal Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soleno Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C602
Record Dates: First submitted 2018-09-27; First posted 2018-10-22 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS; Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OLE DCCR (Experimental): 75 - 525 mg DCCR
  Interventions: Drug: DCCR
- RW DCCR (Experimental): 75 - 525 mg DCCR
  Interventions: Drug: DCCR
- RW Placebo (Placebo Comparator): 75 - 525 mg Placebo for DCCR
  Interventions: Drug: Placebo for DCCR

INTERVENTIONS:
Drug: DCCR — Once daily oral administration of open-label DCCR tablet(s) during the OLE Period
  Arms: OLE DCCR
Drug: DCCR — Once daily oral administration of double-blind (DCCR) tablet(s) during the RW Period
  Arms: RW DCCR
Drug: Placebo for DCCR — Once daily oral administration of double-blind (placebo for DCCR) tablet(s) during the RW Period
  Arms: RW Placebo

SUMMARY:
This is a multi-center, multi-period study with an open-label period followed by a double-blind, placebo-controlled, randomized withdrawal period evaluating the safety and efficacy of DCCR treatment.

DETAILED DESCRIPTION:
115 PWS participants who completed clinical study C601 will be enrolled into the OLE Period. All participants in the Open Label Extension (OLE) Period will receive open-label DCCR. The actual number of participants eligible to enroll in the double-blind, placebo-controlled, randomized withdrawal (RW) period will be limited to those participants taking DCCR in the OLE Period at the time of the RW Period Visit 1 (Baseline/Randomization Visit).The treatment groups in the C602 RW Period are those participants randomized to receive DCCR and those participants randomized to receive Placebo. Participants will be randomized in a 1:1 ratio (DCCR:Placebo).

ELIGIBILITY:
OLE Period Key Inclusion Criteria:

* Successful completion of clinical study C601
* Provide voluntary, written informed consent (parent(s) / legal guardian(s) of patient); provide voluntary, written assent (subjects, as appropriate)

OLE Period Key Exclusion Criteria:

* Positive urine pregnancy test (in females of child-bearing potential) or females who are pregnant or breastfeeding, and/or plan to become pregnant or to breast-feed during or within 90 days after study participation
* Any new disease, condition, or circumstance which would prevent, in the opinion of the Investigator, the patient from completing all study visits and assessments required by the protocol (e.g., an anticipated change of care setting)

RW Period Key Inclusion Criteria:

* Provide voluntary, written informed consent (parent[s] / legal guardian[s] of participant); provide voluntary, written assent (participants, as appropriate); this includes consent for randomization and potential treatment with placebo for up to 16 weeks
* Currently participating in clinical study C602 and complete the OLE End of Treatment Visit procedures

RW Period Key Exclusion Criteria:

* Positive urine pregnancy test (in females of child-bearing potential)
* Females who are pregnant or breastfeeding, and/or plan to become pregnant or to breast-feed during or within 30 days after study participation

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Assess the safety of DCCR by evaluating the incidence and severity of adverse events reported | Baseline to end of OLE (up to 4 years)
  Safety analyses will be conducted in all participants who receive at least one dose of DCCR. Adverse events will be described by type and level of severity.
Change from RW Period Baseline in HQ-CT Total Score | RW Period Baseline to Week 16
  Hyperphagia-related behaviors will be assessed by the hyperphagia questionnaire for clinical trials (HQ-CT), an instrument designed to measure symptoms of food related preoccupations and behaviors. The HQ-CT consists of nine items with responses ranging from 0-4 (best to worst). Scores from 9 items will be summed for a possible total score range of 0-36.

SECONDARY OUTCOMES:
Change from Baseline in HQ-CT Total Score | Baseline to end of OLE (up to 4 years)
  Hyperphagia-related behaviors will be assessed by the hyperphagia questionnaire for clinical trials (HQ-CT), an instrument designed to measure symptoms of food related preoccupations and behaviors. The HQ-CT consists of nine items with responses ranging from 0-4 (best to worst). Scores from 9 items will be summed for a possible total score range of 0-36.
Change in Body Fat Mass | Baseline to end of OLE (up to 4 years)
  Change in Body Fat Mass (kg) using DXA
Clinical Global Impression of Improvement (CGI-I) | RW Period Week 16
  CGI-I is a single statement designed to assess the Investigator's overall perception of change in the subject's condition across the course of the clinical trial. The Investigator provides a response to "Compared to the subject's condition at enrollment, the subject's condition is:" by rating the subject's behavior using a 7-point response scale (best to worst).
Clinical Global Impression of Severity (CGI-S) | RW Period Week 16
  The CGI-S is a single statement designed to assess the Investigator's overall perception of the severity of the participant's illness across the course of the clinical trial. The Investigator provides a response to "Considering your total clinical experience with this particular population, how ill is this participant at this time:" by rating the subject's behavior using a 7-point response scale (best to worst).
Assess the safety of DCCR by evaluating the incidence and severity of adverse events reported | through the end of the RW Period, 16 weeks
  Safety analyses will be conducted in all participants who receive at least one dose of randomized withdrawal study drug. Adverse events will be described by type and level of severity.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (20):
  - University of California, Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida Gainesville, Gainesville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - National Institutes of Health Hatfield Clinical Research Center, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Children's Minnesota, Saint Paul, Minnesota
  - St. Joseph's University Medical Center, Paterson, New Jersey
  - NYU Winthrop Hospital, Mineola, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- United Kingdom (8):
  - The Queen Elizabeth University, Glasgow, Scottland
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, Yorkshire
  - Birmingham Women's and Children's Hospital, Birmingham
  - Fulbourn Hospital, Cambridge
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - Royal London Hospital, London
  - Chelsea and Westminster Hospital, London
  - Hammersmith Hospital, London

REFERENCES:
- [Derived] Strong TV, Miller JL, McCandless SE, Gevers E, Yanovski JA, Matesevac L, Bohonowych J, Ballal S, Yen K, Hirano P, Cowen NM, Bhatnagar A. Behavioral changes in patients with Prader-Willi syndrome receiving diazoxide choline extended-release tablets compared to the PATH for PWS natural history study. J Neurodev Disord. 2024 Apr 26;16(1):22. doi: 10.1186/s11689-024-09536-x. PMID 38671361
- [Derived] Miller JL, Gevers E, Bridges N, Yanovski JA, Salehi P, Obrynba KS, Felner EI, Bird LM, Shoemaker AH, Angulo M, Butler MG, Stevenson D, Goldstone AP, Wilding J, Lah M, Shaikh MG, Littlejohn E, Abuzzahab MJ, Fleischman A, Hirano P, Yen K, Cowen NM, Bhatnagar A; C601/C602 Investigators. Diazoxide choline extended-release tablet in people with Prader-Willi syndrome: results from long-term open-label study. Obesity (Silver Spring). 2024 Feb;32(2):252-261. doi: 10.1002/oby.23928. Epub 2023 Nov 2. PMID 37919617